CLINICAL TRIAL: NCT00750295
Title: An Open Label, Multiple Dose, Time-lagged, Switch Study to Evaluate the Safety, Tolerability and Activity of Escalating SBR759 Doses in Patients With Chronic Kidney Disease on Hemodialysis
Brief Title: A Clinical Study to Evaluate the Safety, Tolerability and Activity of a New Phosphate Binder (SBR759) in Patients With Chronic Kidney Disease on Hemodialysis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSBR759A2101
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2011-08

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic kidney disease,; hemodialysis,; serum phosphorus,; phosphate binders
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — SBR 759

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- 1 (Experimental)
  Interventions: Drug: SBR759
- 2 (Experimental)
  Interventions: Drug: SBR759
- 3 (Experimental)
  Interventions: Drug: SBR759
- 4 (Experimental)
  Interventions: Drug: SBR759
- 5 (Experimental)
  Interventions: Drug: SBR759
- 6 (Experimental)
  Interventions: Drug: SBR759
- 7 (Experimental)
  Interventions: Drug: SBR759

INTERVENTIONS:
Drug: SBR759 — Four weeks of treatment with different doses of SBR759. Patients maintain their prescribed dose of other phosphate binders during the run-in period.
  Arms: 1
Drug: SBR759 — Four weeks of treatment with different doses of SBR759. Patients maintain their prescribed dose of other phosphate binders during the run-in period.
  Arms: 2
Drug: SBR759 — Four weeks of treatment with different doses of SBR759. Patients maintain their prescribed dose of other phosphate binders during the run-in period.
  Arms: 3
Drug: SBR759 — Four weeks of treatment with different doses of SBR759. Patients maintain their prescribed dose of other phosphate binders during the run-in period.
  Arms: 4
Drug: SBR759 — Four weeks of treatment with different doses of SBR759. Patients maintain their prescribed dose of other phosphate binders during the run-in period.
  Arms: 5
Drug: SBR759 — Four weeks of treatment with different doses of SBR759. Patients maintain their prescribed dose of other phosphate binders during the run-in period.
  Arms: 6
Drug: SBR759 — Four weeks of treatment with different doses of SBR759. Patients maintain their prescribed dose of other phosphate binders during the run-in period.
  Arms: 7

SUMMARY:
The primary objective of this study is to assess the safety, tolerability and activity of escalating multiple doses of SBR759 in patients with chronic kidney disease on hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be treated with maintenance hemodialysis and prescribed a phosphate binder.
* A controlled serum phosphorus.
* Constant dose of concomitant medications.
* Women of child bearing potential must be practicing an acceptable form of birth control (i.e. double barrier method - intrauterine device plus condom, spermicidal gel plus condom). All female patients must have a negative pregnancy test at screening in order to be eligible to participate in the study.

Exclusion Criteria:

* Patient has been hospitalized within 30 days prior to screening or has a surgery scheduled during the study.
* Patient has an unstable medical condition, an active infection, active malignancy (except for basal cell carcinoma of the skin), a history of major GI tract surgery, or a history of hemochromatosis.
* Patient is receiving or has received an investigational drug (or is currently using an investigational device) within 30 days prior to screening.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-02; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
In addition to the standard safety assessments (vital signs, ECGs, clinical chemistry and adverse events), serum phosphorus concentration is frequently measured during the study.

SECONDARY OUTCOMES:
Several biomarkers and patient-reported outcomes are assessed at specified time points, before and after treating patients with the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Novartis Investigator Site
Locations (1):
- Novartis Investigator Site, Denver, Colorado, United States

REFERENCES:
- See also: Results for CSBR759A2101 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2639